CLINICAL TRIAL: NCT01508715
Title: Comparison of an Eccentric Exercise Intervention to a Concentric Exercise Intervention in Adults With Subacromial Impingement Syndrome
Brief Title: Comparison of Exercise Interventions in Adults With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16838
Record Dates: First submitted 2012-01-04; First posted 2012-01-12 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Shoulder Impingement Syndrome
Keywords: subacromial; rotator cuff; impingement; physical therapy; eccentric exercise; concentric exercise
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concentric exercise group (Active Comparator): The participants in this group will perform the intervention exercises by actively completing the lifting portion of the resistive shoulder exercises. The physical therapist will then perform the lowering portion of the exercise for the participant.
  Interventions: Other: Shoulder resistive exercise
- Eccentric exercise group (Experimental): The participants in this group will actively perform the lowering portion of the resistive shoulder exercises in the intervention. The physical therapist will perform the lifting portion of the exercise for the participant.
  Interventions: Other: Shoulder resistive exercise

INTERVENTIONS:
Other: Shoulder resistive exercise — Both groups will perform the seated "full can", sidelying internal rotation (IR), sidelying external rotation (ER) with towel roll, supine protraction at 120° of flexion, sidelying horizontal abduction, sidelying abduction, and seated pulley extension using resistance weights in the participant's pain-free shoulder motion. One group will complete only the eccentric portion of the exercise actively, the other will complete only the concentric portion actively. The treating physical therapist will reposition the weights to avoid active resistance occuring in the opposite direction of the desired intervention. Both groups will use 70% of their predicted one repetition maximum (1RM), progressing to 80% with 1RM reassessed and training weight adjusted every two weeks.

SUMMARY:
The purpose of this study is to compare two different physical therapy exercise programs in persons who have shoulder pain in order to determine if they have a different affect on pain level and ability to use the injured shoulder after treatment. Both exercise groups will attend physical therapy for an hour,two to three times a week, for eight weeks. The first two weeks of therapy sessions will involve learning the exercises and testing to determine what weight to use during exercises. One group will perform a traditional therapy exercise program for shoulders using hand weights. The other group will perform a version of the same shoulder exercises but with a different exercise technique. Exercises in both programs are part of the standard of care for shoulder impingement in physical therapy but one program concentrates on the lowering portion of the exercise (eccentrics) while the other emphasizes the lifting portion of the exercise (concentrics). Both groups will perform the same warm-up, stretching, and cool-down exercises. Participants will also be required to perform a daily home exercise program of stretches and range of motion that will take about 20 minutes to complete. Exercise testing will determine the hand weight resistance used by each person during their therapy sessions and re-testing will occur every two weeks to determine any changes in the weight used for the exercises to keep them challenging. Pain level, ability to use the injured arm for daily activities, strength, and amount of movement in the shoulder, will be measured at the start of physical therapy and after five and eight weeks (end of study) of the exercise treatments. A concurrent study investigating the reliability of the shoulder motion and strength measurements used in the larger study will also be performed.

Research hypotheses:

1. Adults with shoulder pain who complete the eccentric progressive resistive exercise intervention will demonstrate significantly greater improvements in the outcome measures at three weeks, earlier in the intervention, than the concentric progressive resistive exercise intervention group.
2. Adults with shoulder pain who perform progressive resistive exercise interventions, regardless of contraction type, will demonstrate significant improvement in the shoulder outcome measures at three and six weeks of intervention.

DETAILED DESCRIPTION:
This study will be a prospective, repeated-measure, randomized clinical trial comparing shoulder outcome measures in adults with SAIS following eccentric or concentric progressive resistance exercise intervention programs. Subjects: 36 persons with SAIS, aged 18 and older, will be recruited from the Texas Health Resources Dallas outpatient rehabilitation department and referring physicians. Procedures: Participants will be randomly assigned to either a concentric or eccentric intervention group. Participants will complete outcome measures for pain intensity, shoulder function, shoulder pain-free active range of motion (AROM) of flexion and scapular plane elevation, and shoulder pain-free strength of external rotation and abduction. Outcomes will be assessed by an investigator blinded to group assignment at baseline and after three and six weeks of intervention. Interventions will consist of supervised exercise sessions three times a week. Exercise progression will follow a standardized and systematic approach. The reliability of the AROM and strength outcome measures will be assessed concurrently using a random subset of six participants from each group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Present with clinical signs of subacromial impingement syndrome
* Have not yet initiated physical or occupational therapy treatment

Exclusion Criteria:

* Previous shoulder, cervical, or thoracic surgery.
* History of shoulder fracture, dislocation, labral tear, or full thickness rotator cuff tear
* Treatment for neoplasm in the last year
* Rheumatic disease
* Adhesive capsulitis
* Shoulder pain currently rated greater than or equal to 8/10 on the NPRS
* Cardiac, neurological, or musculoskeletal condition that precludes ability to perform upper extremity resisted exercise
* Pregnancy
* inability to understand spoken or written English
* Inability to arrange transport to evaluation or treatment sessions or not planning to stay in the area long enough to complete study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder function | baseline, after 3 weeks and 6 weeks of intervention
  Measured by change in numeric pain rating scale (NPRS)score for shoulder pain, change in disabilities of the arm, shoulder, and hand (DASH) self-report of function score, change in shoulder abduction and external rotation strength assessed with a hand-held dynamometer, and change in shoulder flexion and scapular plane elevation pain-free range of motion assessed with a digital inclinometer.

SECONDARY OUTCOMES:
Intratester reliability | over course of study
  A subset of participants will be tested for strength and range of motion outcomes twice at each time frame by the same examiner in order to analyze intratester reliability of the testing protocols using Intraclass Correlation Coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Christiana L Blume, PT, PhD, OCS, Principal Investigator — Texas Woman's University, Texas Health Resources, Dallas
Locations (1):
- Texas Health Resources, Presbyterian Hospital, Dallas, Texas, United States